CLINICAL TRIAL: NCT03135197
Title: German Observational Multicenter Study of Patients With Fabry Disease Under Chaperone Therapy With Migalastat-HCl.
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: Fabry_Migalastat
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migalastat: Migalastat administered according to SmPC

SUMMARY:
The objective of the study is to document long term data on treatment with Migalastat under "real world" conditions. The selection of patients is based on the SmPC/Fachinformation. The study duration/patient will be 2 years.

DETAILED DESCRIPTION:
Phase 3 data should be confirmed in this study with long-term data.

* LVMI is expected to remain stable or to be ameliorated over an average of 24 months treatment duration. The LVMI reduction observed in patients followed up to 24 months is expected to be significantly reduced with a mean change of -6.6 g/m2 (-11.0, -2.1, 95% CI).
* eGFR [CKD-EPI] is expected to remain stable over an average of 24 months treatment duration. The long-term effect of Migalastat on eGFR is expected to be comparable to the decline over time in healthy adults. The annualized rate of change over this period is expected to be ≤1 mL/min/1.73 m2 in females and ≤3 mL/min/1.73 m2 in males.
* Significant reduction is expected in plasma lyso-Gb3 concentration at month 6, month 12 and month 24 following treatment with Migalastat.
* ERT-naïve patients treated with Migalastat are expected to show an improvement of GI symptoms (diarrhea) over 24 months.
* No progression of White Matter Lesions (WML) during treatment duration is expected.
* No higher frequency of stroke/transient cerebral ischemia during treatment duration is expected.
* Severity of neuropathic pain is expected to remain stable or to improve during treatment duration.
* Dosing/amount of symptomatic medications of neuropathic symptoms is expected to decrease during treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 16 to 74 years, diagnosed with Fabry disease.
* Amenable GLA mutation.
* Treatment with Migalastat (initiation of therapy according to recommendations for initiation and cessation of enzyme replacement therapy in patients with Fabry disease: the European Fabry Working Group consensus document. Biegstraaten et al, Orphanet J Rare Dis. 2015;10:36. AWMF-Leitlinien Morbus Fabry, Diagnose und Therapie, Registernummer 030-134).

The following Inclusion criteria refer to the time of Migalastat initiation (T0):

* ERT naïve (patients with signs of organ involvement (kidney, heart and/or CNS signs) to be considered for ERT following the European Consensus Guidelines on ERT (Biegstraaten et al 2015) or patients with neuropathic pain not controlled with pain medication or patients with GI symptoms not relieved with standard medication or ERT switch patients (under ERT for ≥12 months).
* Estimated GFR (eGFR, CKD-EPI formula) at screening ≥30 ml/min/1.73 m2
* Subjects taking no ACE inhibitors, ARBs, or renin inhibitors or are on a stable dose for at least 4 weeks before screening.
* Subjects taking no analgesics/antidepressants or are on a stable dose for at least 4 weeks before screening.

Exclusion Criteria:

* Patient has a non-amenable GLA mutation or the mutation A143T or D313Y (for verification of amenable mutations please refer to: www.GalafoldAmenablityTable.com or to the "Fachinformation").
* Patient is unwilling to give informed consent.
* Patient is unable to comply with the clinical protocol.
* Patients on co-medication: Galafold plus Enzyme Replacement Therapy (ERT)
* Pregnant or breast feeding women.

The following Exclusion criteria refer to the time of Migalastat initiation (T0):

* Patients on dialysis
* Patient has a clinically significant organ disease (e.g. cancer in the past 5 years) that in the opinion of the investigator would preclude participation in the trial.
* Patients with a history of organ transplantation.

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: At therapy initiation adult male and female patients with FD will be identified, whose GLA mutations are amenable for a stimulation with Migalastat-HCl, and will be treated with Migalastat-HCl at the recommended dose continuously for 24 months according to the manufacturers' instructions (SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
LVMI | two years
  Primary endpoint of the observational study is the change in left ventricular mass index (LVMI) over two years.

SECONDARY OUTCOMES:
GFR | 24 months
  Change in GFR over 24 months
Cerebral ischemia or stroke. | 24 months
  Incidence of transient/manifest cerebral ischemia or stroke over 24 months.
Neuropathic Pain (GCPS) | 24 months
  Change in severity of neuropathic pain measured by Graded Chronic Pain Scale (GCPS)
Neuropathic Pain (NPSI) | 24 months
  Change in severity of neuropathic pain measured by Neuropathic Pain Symptom Inventory (NPSI) Score (items are quantified on a (0-10) numerical scale).
Fabry Disease Severity (MSSI) | 24 months
  Change in disease severity measured by Mainz Severity Score Index (MSSI)
Fabry Disease Severity (DS3) | 24 months
  Change in disease severity measured by the Disease Severity Scoring System (DS3)
Lyso-Gb3 | 24 months
  Change in Lyso-Gb3
White Matter Lesion load | 24 months
  Change of White Matter Lesion load (quantified by WML volumetry [ml]).
Cerebral microbleeds/hemorrhagic lesions. | 24 months
  Stabilization of cerebral microbleeds/hemorrhagic lesions.
Gastrointestinal symptoms | 24 months
  Change in gastrointestinal symptoms (gastrointestinal symptoms rating scale, GSRS).
Quality of life (SF-36) | 24 months
  Change in quality of life (Short Form (SF-36) Health Survey: 36-item, patient-reported survey of patient health).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Brand, Prof., Principal Investigator — University Hospital Muenster
Locations (1):
- Universtiy Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No